CLINICAL TRIAL: NCT02588846
Title: Phase I Feasibility Study of Accounting for Relative Motion of Multiple Targets in Prostate Cancer Radiotherapy Using Realtime Multi-leaf Collimator Adaptation and Kilovoltage (kV) Intrafraction Monitoring
Brief Title: Multi-target Tracking in Prostate Radiotherapy Using MLC and KIM
Acronym: KOALA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no resources to run the trial
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Professor Thomas Eade, Head of Research, Royal North Shore Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Multi-target tracking
Record Dates: First submitted 2015-07-14; First posted 2015-10-28 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: Prostate; Radiotherapy; IGRT; VMAT; Image-guided radiation therapy; Volumetric modulated arc therapy; Adaptive radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients receive the intervention for comparison against retrospective matched cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1: Optimise nodal treatment margin (Experimental): During Stage 1: Optimise nodal treatment margin, Combined real-time use of 'Multi-Leaf Collimator Adaptation' and 'kV Intrafraction Monitoring' will be used to reshape the radiation beam in real-time. The nodal target position stability will be evaluated by the cone beam computed tomography (CBCT) imaging before and after each treatment session for the first 10 patients.
  Interventions: Device: Combined real-time use of 'Multi-Leaf Collimator Adaptation' and 'kV Intrafraction Monitoring'
- Stage 2: Use treatment margin (Experimental): During Stage 2: Use treatment margin, Combined real-time use of 'Multi-Leaf Collimator Adaptation' and 'kV Intrafraction Monitoring' will be used to reshape the radiation beam in real-time. At the same time, multi-leaf collimator (MLC) tracking will be used to reshape the radiation beam in real-time using the margin size determined in Stage 1.
  Interventions: Device: Combined real-time use of 'Multi-Leaf Collimator Adaptation' and 'kV Intrafraction Monitoring'

INTERVENTIONS:
Device: Combined real-time use of 'Multi-Leaf Collimator Adaptation' and 'kV Intrafraction Monitoring' — This intervention uses the simultaneous combined use of two technologies: 'Multi-Leaf Collimator Adaptation' and 'kV Intrafraction Monitoring'. kV Intrafraction Monitoring (KIM) measures the motion of tissues targeted for radiotherapy in real time using kV imaging.The multi-leaf collimator (MLC) reshapes the radiation beam to maximise dose to the target tissue and minimise dose to the surrounding healthy tissue. Combining KIM and MLC allows the shaped radiation beam to follow the moving target (the prostate) while remaining fixed on a stationary target (lymph nodes) that are also being treated at the same time.
  Other Names: MLC; KIM

SUMMARY:
Assessing the feasibility of implementing real-time multi-leaf collimator (MLC) tracking to account for the relative motion of the moving prostate tumour target and the static pelvic nodal target for high-risk prostate cancer patients. The capability of tracking for the relative motion of multiple targets will ensure that all the treatment targets receive correct dose as prescribed by the doctor and minimise side effects to the critical organs.

DETAILED DESCRIPTION:
This study will assess the feasibility of implementing real-time multi-leaf collimator (MLC) tracking to account for the relative motion of the moving prostate tumour target and the static pelvic nodal target for high-risk prostate cancer patients. The capability of tracking for the relative motion of multiple targets will ensure that all the treatment targets receive correct dose as prescribed by the doctor and minimising side effects to the critical organs.

During radiation treatment, the prostate position will be monitored in real time using the KIM technology. The nodal target will be imaged before and after each treatment to evaluate the nodal treatment margin. The MLC tracking is implemented by recalculating the radiation beam shape fit for the moved prostate and static nodal targets and sending the adjusted MLC leaf positions to the treatment delivery system. The actually delivered dose to the patient will be calculated after the treatment and compared to the dose without MLC tracking to assess the treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing definitive external beam radiotherapy at Northern Sydney Cancer Centre
* Patients histologically proven prostate adenocarcinoma
* PSA obtained within 3 months prior to enrolment
* Pelvic lymph nodes are included for treatment for patients at stage T1c-T3b with Gleason 8-10 or prostate-specific antigen (PSA) > 20 ng/ml or pelvic lymph node positivity on conventional imaging or prostate-specific membrane antigen (PSMA) scans.
* Patient must be able to have gold fiducial markers placed in the prostate
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document.
* Prostate dimension that allows leaf span with tracking margin of ±8mm

Exclusion Criteria:

* Patients with artificial Hip(s), lumbar spinal surgical rods or other large metallic pelvic implants
* Patient's dimensions >40cm as measured at the level of the prostate
* Patients with overlapping implanted gold fiducials in x-ray imaging

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Software or mechanical failure | The treatment period (2-9 weeks)
  The percentage of fractions delivered without software or mechanical failure

SECONDARY OUTCOMES:
Geometric accuracy | The treatment period (2-9 weeks)
  The geometric accuracy of the beam shape, determined by comparing the ideal beam shape with the actual beam shape.
Prostate motion trajectory | Treatment period (2-9 weeks)
  Prostate motion trajectory measured by KIM.
Dosimetric accuracy | Treatment period (2-9 weeks)
  The estimated dose distributions will be compared to the original plan using the dose reconstruction method18 based on the prostate motion trajectory and the logged MLC positions (beam shapes).
Acute toxicity | Treatment period (2-9 weeks) plus 3 months
  Toxicity during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eade, MBBS, RANZCR, Principal Investigator — Director of Research, Senior Staff Specialist
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Share for research purposes with interested parties.